CLINICAL TRIAL: NCT07344857
Title: Impact of a Prenatal Pilates Program Continued Until Childbirth on Postpartum Ligamentous Recovery: a Longitudinal Follow-up of a Randomized Controlled Trial
Brief Title: Prenatal Pilates and Postpartum Ligamentous Laxity
Status: Completed | Type: Observational
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, Selcan Suicmez, Research Asst., Ankara Medipol University
Other Study IDs: AnkaraMedipolU-FTR-2025-223
Record Dates: First submitted 2026-01-08; First posted 2026-01-15 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Laxity of Ligament; Pregnancy; Pilates Exercise
MeSH Terms: conditions — Joint Instability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pilates Group: Participants in the Pilates group attended supervised 60-minute sessions twice weekly for eight weeks, led by a certified physiotherapist trained by the Australian Institute of Pilates and Physiotherapy.
- Control Group: The control group received standard prenatal care and ergonomic advice, and did not participate in any exercise training.

SUMMARY:
Pregnancy induces hormonal and biomechanical adaptations that increase ligamentous laxity, which may persist into the postpartum period and contribute to joint instability, pain, and functional limitations. Although prenatal Pilates has been shown to prevent the progression of ligamentous laxity during pregnancy, its effects on postpartum musculoskeletal recovery remain unclear. This longitudinal follow-up of a randomized controlled trial evaluated ligamentous recovery at 6 weeks postpartum in women who participated in a structured prenatal Pilates program continued until childbirth, compared with women receiving standard prenatal care. Postpartum ligamentous laxity, generalized joint hypermobility, and activity limitations related to pelvic girdle pain were assessed using objective and clinical measures. The study aimed to determine whether prenatal Pilates facilitates early postpartum ligamentous recovery and supports functional outcomes during the early postpartum period.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-35 years
* In the 6th week of post-partum
* Voluntary participation in the study

Exclusion Criteria:

* Cardiovascular or pulmonary diseases
* Prior participation in structured physical activity programs

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Study Population: The study population consisted of postpartum women aged 18-35 years who were 6th week after delivery and who voluntarily agreed to participate in the study. Women with known cardiovascular or pulmonary diseases, and those who had participated in structured physical activity programs prior to enrollment were excluded. These criteria were applied to ensure a homogeneous sample and to minimize potential confounding factors related to pre-existing health conditions or prior exercise exposure.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Ligament laxity | 10 minutes
  The anterior tibial translation of the knee will be considered as representative of the anterior laxity of the knee of women measured with an arthrometer ® (bilateral examination repeated 3 times on each knee).The degree of laxity will be evaluated thanks to the international classification IKDC.

SECONDARY OUTCOMES:
Generalized joint hypermobility | 2 minutes
  Generalized joint hypermobility (GJH) was assessed using the Beighton scoring system, which consists of five bilateral and unilateral maneuvers. Each positive test scored one point, with a maximum score of 9. A score of ≥5 indicated GJH.
Physical activity level | 7 days
  Participants' physical activity was monitored using the Omron HJ-321-E pedometer (Omron Healthcare, Japan), which detects vertical oscillations and stores up to seven days of data.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Medipol University, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No